CLINICAL TRIAL: NCT02847312
Title: Chronic Cardiovascular and Gut-bacteria Effects of Phenolic Rich Oats in Adults With Above Average Blood Pressure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Reading (Other)
Collaborators: PepsiCo, Inc. (Industry); Rothamsted Research (Unknown); Biotechnology and Biological Sciences Research Council (Other)
Responsible Party: Principal Investigator, Jeremy Paul Edward Spencer, Professor, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Prograin3
Record Dates: First submitted 2016-07-25; First posted 2016-07-28 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Healthy
Keywords: Oat; Phenolic acid; Avenanthramide; FMD; LDI; Gut microbiota; Blood Pressure; Renin Angiotensin; Nitric Oxide
MeSH Terms: conditions — Gyrate Atrophy | interventions — phenolic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- High avenanthramide, phenolic acid (Active Comparator): 66.8g Pepsico Oatmeal + 60g Oat cake
  Interventions: Other: High avenanthramide, phenolic acid
- Low avenanthramide, medium phenolic acid (Active Comparator): 17g Oatwell + 63.6g Cream of Rice + 60g Melba Toast
  Interventions: Other: Low avenanthramide, medium phenolic acid
- Control (Placebo Comparator): 69.8g Cream of Rice + 8.1g Cellulose + 4.8g Pectin + 60g Melba Toast
  Interventions: Other: Control

INTERVENTIONS:
Other: High avenanthramide, phenolic acid — High avenanthramide and high phenolic acid, matched with energy and insoluable fibre.
  Arms: High avenanthramide, phenolic acid
Other: Low avenanthramide, medium phenolic acid — Low avenanthramide and moderate phenolic acid, matched with energy and insoluable fibre.
  Arms: Low avenanthramide, medium phenolic acid
Other: Control — Control are matched with energy and insoluable fibre.
  Arms: Control

SUMMARY:
In this proposed human trial, the investigators aim to establish whether 4 weeks of daily consumption of beta-glucan matched meals providing either a high dose or a moderate dose of oat avenanthramides and phenolic acids leads to dose-dependent chronic improvements in markers of CVD risk and gut health relative to an energy matched control intervention in healthy adults with above average blood pressure.

DETAILED DESCRIPTION:
* To investigate the chronic effects of daily intake of oat products on flow mediated dilatation of the brachial artery (FMD; primary endpoint), microvascular endothelial function (measured by laser Doppler iontophoresis), pulse wave analysis, gut microbiota diversity, 24h blood pressure, activity of the renin angiotensin system, markers related to cellular production of nitric oxide and reactive oxygen species, inflammatory cytokines, and further potentially emerging biochemical markers of CVD risk.
* To establish if phenolic acids and avenanthramides from oat products exert cardiovascular and microbial effects in a dose dependent manner.
* To measure urinary and fecal excretion of avenanthramide and phenolic acid metabolites.

To explore correlations between bacterial population changes and CVD risk markers.

ELIGIBILITY:
Inclusion Criteria:

* Above average blood pressure (i.e. systolic 120-159 mmHg and diastolic 75-99 mmHg)

Exclusion Criteria:

* Abnormal biochemical, haematological results as assessed at health screening
* Hypertension (i.e. SBP/DBP ≥160/100 mm Hg)
* BMI >35
* Current smoker or ex-smoker ceasing <3 months ago
* Past or existing medical history of vascular disease, diabetes, hepatic, renal, haematological, neurological, thyroidal disease or cancer
* Prescribed or taking lipid lowering, antihypertensive, vasoactive (e.g. Viagra), anti-inflammatory, antibiotic or antidepressant medication
* Allergies to whole grains
* Parallel participation in another research project
* Having flu vaccination or antibiotics within 3 months of trial start
* Chronic constipation, diarrhea or other chronic gastrointestinal complaint
* On a weight reduction regime or taking food, probiotics or prebiotics supplements or laxative within 3 months of trial start
* Performing high level of physical activity (i.e. ≥150min aerobic exercise/week)
* Consumption of ≥21 units of alcohol/week
* Females who are breast-feeding, may be pregnant, lactating or, if of reproductive age and not using a reliable form of contraception (including abstinence)

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Flow mediated dilatation | 20 weeks
  Technique to assess the flexibility of teh endothelium in larger peripheral blood vessels, magnitude of increase in percentage from baseline to after 4 weeks treatment.

SECONDARY OUTCOMES:
Laser Doppler Iontophoresis | 20 weeks
  Magnitude of increase from Baseline to 4weeks treatment
Gut microbiota changes | 22 weeks
  Gut microbiota diversity and relative abduance change from Baseline to 4weeks treatment
Plasma nitric oxide analysis | 22 weeks
  Concentration of nitric oxide in nmol from Baseline to 4weeks treatment
NADPH oxidase activity in neutrophil blood cells | 22 weeks
  NADPH oxidase activity will be calculated as the difference between values obtained in PMA from Baseline to 4weeks treatment
Inflammatory markers | 22 weeks
  Inflammatory marker levels change from Baseline to 4weeks treatment
Renin activity | 22 weeks
  Renin activity in ng/(mL*hour)
Plasma microparticles | 22 weeks
  Microparticles in counts/uL
Urine and plasma metabolomic footprint using NMR | 22 weeks

OTHER OUTCOMES:
Plasma glucose | 22 weeks
  Glucose concentration in mmol/L
Plasma insulin | 22 weeks
  Insulin concentration in uU/mL
Plasma lipids | 22 weeks
  Plasma lipid concentration in mmol/L
Faecal water metabolites | 22 weeks
  Metabolites in mikrogram/L

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy P Spencer, Professor, Principal Investigator — University of Reading
Locations (1):
- Hugh Sinclair Unit of Human Nutrition, Reading, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Publish